CLINICAL TRIAL: NCT06871800
Title: Evaluation of Predictive Circulating Biomarkers for Rehabilitation Recovery in Ischemic and Haemorrhagic Stroke Patients: From Lacunar Stroke to Vascular Severe Brain Injury
Brief Title: Blood Extracellular Vesicles as Predictive Recovery Biomarker After Stroke and Brain Injury
Acronym: PRISMA
Status: Recruiting | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Other Study IDs: PRISMA; CET 65/24 (Other: CET Lombardia 4, Milan, Italy)
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Stroke; Vascular Severe Brain Injury; Rehabilitation
Keywords: stroke; brain injury; biomarkers; biosensor; response to treatment
MeSH Terms: conditions — Stroke; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples used for extracellular vesicles isolation. DNA content will be not considered
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Stroke patients: 30 post-stroke patients will be enrolled at IRCCS S. Maria Nascente (Milan), S. Maria ai Colli (Turin) and IRCCS Don Gnocchi (Florence) of Fondazione Don Gnocchi.
  Interventions: Other: blood withdrawal
- Patients with vascular severe brain injury: 30 patients with vascular severe brain injury (vSBI) will be enrolled at IRCCS S. Maria Nascente (Milan), and S. Maria ai Colli (Turin) of Fondazione Don Gnocchi.

INTERVENTIONS:
Other: blood withdrawal — 10 ml of blood, two 5 ml tubes suitable for serum isolation. Blood collection will be done at admission in the rehabilitation department (T0), after completing 50% of their rehabilitation program (T1), and at discharge (T2)
  Groups: Stroke patients

SUMMARY:
The rehabilitation outcome and recovery, in people after stroke or with vascular severe brain injury(vSBI), are difficult to predict. Moreover, the clinical management of patients during hospitalization is problematic due to complex clinical conditions and complications, e.g. healthcare-associated infections(HAIs). Today we still lack early objective biomarkers that could predict the patient's trajectory at admission. Extracellular vesicles are nanoparticles naturally released by cells in physiological and pathological conditions. As important actors of cellular communication between different organs and body districts, EVs are currently under investigation as an informative tool able to reflect the clinical conditions of patients. Using an optimized Surface Plasmon Resonance imaging (SPRi) based biosensor, our main objective is to assess the predictive capacity of biomarkers associated to blood-derived extracellular vesicles for anticipating patients' recovery after stroke and vSBI. If successful, the project will 1) demonstrate the ability of the SPRi biosensor to reveal differences in the relative amount of specific cell-derived EV subpopulations and their molecular cargo during disease progression and rehabilitation-induced recovery, 2) verify the impact of HAI on patients' response, 3) perform a patient's stratification to personalize the rehabilitation protocol.

DETAILED DESCRIPTION:
OBJECTIVE: The main objective of the present project is to assess the predictive capacity of biomarkers associated to extracellular vesicles (EVs) for anticipating patients' recovery after stroke and vSBI.

The characterization by SPRi of different cell-derived families of EVs (endothelium, neurons, microglia, muscle, and neutrophil) will allow to evaluate the activation status of the processes of neuroinflammation, neuronal regeneration, and angiogenesis to provide a picture of the mechanisms of response to the damage taking place in the brain of patients and enhanced by the rehabilitation treatment. The selected markers are expected to be released in the brain, but they can be monitored in the periphery taking advantage of the ability of EVs to cross the blood-brain barrier.

Due to the weight of HAIs on patients' prognosis, inflammation and infections will represent the main covariate of the analysis in the search for predictive rehabilitation biomarkers.

Specific objectives are as follows:

1. Evaluation of the SPRi biosensor's ability to detect EV-associated biomarkers correlating with stroke severity.
2. Evaluation of the ability of EV-associated biomarkers to represent a recovery biomarker by their changes according to the patient's outcome.
3. Evaluation of the ability of EV-associated biomarkers to identify infection-prone patients to help develop valuable prevention strategies for infections.

These data will be correlated with the outcome of the rehabilitation evaluated with specific functional and neurological scales that allow accurate profiling of the patient and the evaluation of functional recovery.

IMPACT: The primary impact of the present project is the clinical management of the neurorehabilitation department for stroke and vSBI patients. The identification of measurable biomarkers that could predict the response to rehabilitation of patients and group them into responders or non-responders would significantly modify the everyday activity of physiatrists. In the long term, patients will take advantage of a personalized treatment that will lead to optimal recovery. Optimal intervention and recovery imply amelioration of the quality of life of patients and their families and reduced time and costs of the intervention.

SAMPLE COLLECTION: 30 stroke patients will be recruited at IRCCS S. Maria Nascente (Milan), S. Maria ai Colli (Turin), and IRCCS Don Gnocchi (Florence), while 30 subjects with vSBI will be recruited at IRCCS S. Maria Nascente (Milan) and S. Maria ai Colli (Turin) of Fondazione Don Gnocchi. Recruited patients will undergo blood withdrawal (10 ml of blood for serum separation) at 3 time points: at admission in the rehabilitation department (T0), after completing 50% of their rehabilitation program (T1), and at discharge (T2).

EV ISOLATION: EVs isolation will be perfomed at the Laboratory of Nanomedicine and Clinical Biophotonics of IRCCS S. Maria Nascente (Milan). EVs will be isolated from serum by size exclusion chromatography. To evaluate the size distribution and the concentration of the isolated EVs, the Nanoparticle Tracking Analysis (NTA) will be carried out. Reported markers of small EVs will be evaluated by Western blot to verify the successful isolation.

SPRi BIOSENSOR: The functionalization of the SPRi chip will be optimized for marker of endothelial EVs (CD31), neuronal EVs (CD171/L1CAM), microglia Evs (IB4), muscle EVs (Irisin), and neutrophil EVs (CD15 or CD66b).

Correlation analysis will be performed between SPRi-data and clinical measures at admission (T0), T1 and T2, separately. Correlation analysis will be performed also between the biomolecular markers measured at T0 and the change scores obtained from clinical assessments to test their ability to predict the outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Disability deriving from first ischemic or haemorrhagic stroke detected by MRI or CT scan
* Time from stroke onset or rehabilitation admission less than 1 month (for stroke) 3 months (for vSBI)
* Need of inward rehabilitation
* Signed informed consent by patient or legal representative

Exclusion Criteria:

* Subarachnoid haemorrhage
* Cerebral venous thrombosis
* Other previous neurological or psychiatric conditions
* Autoimmune diseases
* Previous severe and chronic infections conditions (e.g. tuberculosis, HIV/AIDS)
* Neoplasms or other malignant conditions
* Immunomodulatory medications (immunosuppressants).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized at Fondazione Don Gnocchi (IRCCS S. Maria Nascente/Milan, S. Maria ai Colli/Turin, and IRCCS Don Gnocchi/Florence) after stroke injury or with vascular severe brain injury and undergoing an intensive rehabilitation program.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in modified Barthel index after rehabilitation | From admission in the rehabilitation department (T0) to discharge (T2; max 2 months from enrollment)
  Modified Barthel index (Shah et al., 1989) validated in the literature and already proposed in the PMIC 2020 and PMGCA 2020 by SIMFER, will be used for accurate patient profiling and assessment of functional recovery (for all groups).

SECONDARY OUTCOMES:
Extracellular vesicles characterization by SPRi | From admission in the rehabilitation department (T0) to discharge (T2; max 2 months from enrollment)
  Changes in biomarkers expression associated to EVs (CD9, CD31, CD171, IB4, CD11b, IRISIN, CD15/CD66b) from serum, by SPRi biosensor. Changes between baseline (T0) and samples at T1 (15-20days after T0) and T2 (after rehabilitation, max 2 months) will be evaluated (for all groups).
Change in National Institute of Health Stroke Scale (NIHSS) (for stroke) | From admission in the rehabilitation department (T0) to discharge (T2; max 2 months from enrollment)
  NIHSS scale (Brott et al. 1989) , validated in the literature and already proposed in the PMIC 2020 by SIMFER, will be used for accurate patient profiling and assessment of functional recovery .
  Changes between baseline (T0) and samples at T1 (15-20days after T0) and T2 (after rehabilitation, max 2 months) will be evaluated (for stroke).
Change in Coma Recovery Scale (for vSBI) | From admission in the rehabilitation department (T0) to discharge (T2; max 2 months from enrollment)
  Coma Recovery Scale (Giacino & Kalmar, 2004) validated in the literature and already proposed in the PMGCA 2020 by SIMFER, will be used for accurate patient profiling and assessment of functional recovery. Changes between baseline (T0) and samples at T1 (15-20days after T0) and T2 (after rehabilitation, max 2 months) will be evaluated (for vSBI).
Change in Level of Cognitive Functioning (LCF) (for vSBI) | From admission in the rehabilitation department (T0) to discharge (T2; max 2 months from enrollment)
  Level of Cognitive Functioning (Francesco Lombardi, 2002) validated in the literature and already proposed in the PMGCA 2020 by SIMFER, will be used for accurate patient profiling and assessment of functional recovery.
  Changes between baseline (T0) and samples at T1 (15-20days after T0) and T2 (after rehabilitation, max 2 months) will be evaluated (for vSBI).
Change in Glasgow Outcome Scale - Extended (GOSE) (for vSBI) | From admission in the rehabilitation department (T0) to discharge (T2; max 2 months from enrollment)
  Glasgow Outcome Scale Extended (J Neurotrauma, 1998) validated in the literature and already proposed in the PMGCA 2020 by SIMFER, will be used for accurate patient profiling and assessment of functional recovery.
  Changes between baseline (T0) and samples at T1 (15-20days after T0) and T2 (after rehabilitation, max 2 months) will be evaluated (for vSBI).
Change in Rehabilitation Complexity Scale (for all groups) | From admission in the rehabilitation department (T0) to discharge (T2; max 2 months from enrollment)
  Rehabilitation Complexity Scale (Lynne Turner-Stokes, 2007) validated in the literature and already proposed in the PMGCA 2020 by SIMFER, will be used for accurate patient profiling and assessment of functional recovery.
  Changes between baseline (T0) and samples at T1 (15-20days after T0) and T2 (after rehabilitation, max 2 months) will be evaluated (for all groups).
Change in Mini Mental State Evaluation (MMSE) (for stroke) | From admission in the rehabilitation department (T0) to discharge (T2; max 2 months from enrollment)
  MMSE (T Nissen, 1989) validated in the literature and already proposed in the PMIC 2020 and PMGCA 2020 by SIMFER, will be used for accurate patient profiling and assessment of functional recovery.
  Changes between baseline (T0) and samples at T1 (15-20days after T0) and T2 (after rehabilitation, max 2 months) will be evaluated (for stroke).
Change in Modified RANKIN scale (mRS) (for all groups) | From admission in the rehabilitation department (T0) to discharge (T2; max 2 months from enrollment)
  Modified RANKIN scale (G Popa, 1992) validated in the literature and already proposed in the PMIC 2020 and PMGCA 2020 by SIMFER, will be used for accurate patient profiling and assessment of functional recovery.
  Changes between baseline (T0) and samples at T1 (15-20days after T0) and T2 (after rehabilitation, max 2 months) will be evaluated (for all groups).

CONTACTS AND LOCATIONS:
Overall Officials: Alice Gualerzi, PhD, Principal Investigator — Fondazione Don Carlo Gnocchi, Laboratory of Nanomedicine and Clinical Biophotonics
Locations (3):
- Italy (3):
  - IRCCS "Don Gnocchi", Fondazione Don Gnocchi Onlus, Florence
  - IRCCS "S. Maria Nascente", Fondazione Don Gnocchi Onlus, Milan
  - "S. Maria ai Colli - Presidio Ausiliatrice", Fondazione Don Gnocchi Onlus, Torino

IPD SHARING:
Plan to Share IPD: No
All personal data will be pseudoanonimized upon collection and reported in publications and scientific presentations only as anonymous and/or aggregated data that do not allow to trace the identity of the involved subjects.

REFERENCES:
- [Background] Gualerzi A, Picciolini S, Roda F, Bedoni M. Extracellular Vesicles in Regeneration and Rehabilitation Recovery after Stroke. Biology (Basel). 2021 Aug 30;10(9):843. doi: 10.3390/biology10090843. PMID 34571720
- [Background] Picciolini S, Gualerzi A, Carlomagno C, Cabinio M, Sorrentino S, Baglio F, Bedoni M. An SPRi-based biosensor pilot study: Analysis of multiple circulating extracellular vesicles and hippocampal volume in Alzheimer's disease. J Pharm Biomed Anal. 2021 Jan 5;192:113649. doi: 10.1016/j.jpba.2020.113649. Epub 2020 Sep 23. PMID 33038641
- [Background] Picciolini S, Gualerzi A, Vanna R, Sguassero A, Gramatica F, Bedoni M, Masserini M, Morasso C. Detection and Characterization of Different Brain-Derived Subpopulations of Plasma Exosomes by Surface Plasmon Resonance Imaging. Anal Chem. 2018 Aug 7;90(15):8873-8880. doi: 10.1021/acs.analchem.8b00941. Epub 2018 Jul 17. PMID 29972017
- [Background] Picciolini S, Mangolini V, Roda F, Montesano A, Arnaboldi F, Liuzzi P, Mannini A, Bedoni M, Gualerzi A. Multiplexing Biosensor for the Detection of Extracellular Vesicles as Biomarkers of Tissue Damage and Recovery after Ischemic Stroke. Int J Mol Sci. 2023 Apr 27;24(9):7937. doi: 10.3390/ijms24097937. PMID 37175644
- See also: Laboratory of Nanomedicine and Clinical Biophotonics, Fondazione Don Carlo Gnocchi — http://www.labion.eu